CLINICAL TRIAL: NCT04707807
Title: Effects of Nightshift Work and Sleep Disturbances on Erectile Function, Serum Testosterone Levels, Nocturia
Brief Title: Effects of Nightshift Work and Sleep Disturbances on Erectile Function
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istanbul Medipol University Hospital (Other)
Collaborators: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, gokhan calik, Assistant professor, Istanbul Medipol University Hospital
Other Study IDs: MedipolUrology
Record Dates: First submitted 2021-01-12; First posted 2021-01-13 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Erectile Dysfunction, Nocturia, Short Term Insomnia, Obstructive Sleep Apnea
MeSH Terms: conditions — Erectile Dysfunction; Nocturia; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Nightshift workers
  Interventions: Diagnostic Test: IIEF-5
- Non-nightshift workers
  Interventions: Diagnostic Test: IIEF-5

INTERVENTIONS:
Diagnostic Test: IIEF-5 — IIEF-15 form will be filled out by all participants

SUMMARY:
We aim to observe the unwanted effects of nightshift work and short term insomnia on erectile function of men aged between 25 to 60 years. We will also compare the levels of serum testosterone in the target group and compare it with the ones who don't work in hightshifts.

ELIGIBILITY:
Inclusion Criteria:

* Suffering from erectile dysfunction
* Mainly psychogenic ED
* Employed

Exclusion Criteria:

* Patients with major organic causes erectile dysfunction (Radical pelvic surgery/radiation therapy, uncontrolled diabetis mellitus, uncontrolled hypertension, New York Heart Association Class 3-4 heart failure, acute coronary syndrome within 3 months, dyslipidemia)
* NEET(Not in employment, education, training) patients

Ages: 25 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: We aim to enroll mainly working class men in our study. So we are going to be able to compare the erectile function status daytime workers with nightshifters. Unemployed, retired and students will be excluded form the study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-11-20 (Actual); Primary Completion 2021-05-20 (Estimated); Study Completion 2021-11-20 (Estimated)

PRIMARY OUTCOMES:
Erectile dysfunction | 3-6 months
  Decreased scores of IIEF-5

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Istanbul Medipol University Hospital, Bağcılar, Istanbul
  - Cemil Tascioglu Cith Hospital, Istanbul, Sisli

IPD SHARING:
Plan to Share IPD: No